CLINICAL TRIAL: NCT05156827
Title: A Phase 2 Double-blind, Randomized, Multi-center, Parallel-group Study to Assess the Efficacy, Safety, and Pharmacokinetics of TB006 in Patients With Acute Ischemic Stroke
Brief Title: A Study to Assess the Efficacy, Safety, and Pharmacokinetics of TB006 in Participants With Acute Ischemic Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TB006AIS2103
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke (AIS); TB006; stroke; efficacy; safety; pharmacokinetics; ischemia
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia | interventions — TB006

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TB006 (Experimental): Participants will receive intravenous (IV) 3 infusions of 4000 milligrams (mg) TB006, one every 28 days (Q28D).
  Interventions: Drug: TB006
- Placebo (Placebo Comparator): Participants will receive an IV infusion of normal saline 500 milliliters (mL) Q28D.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TB006 — TB006 diluted in normal saline, administered through IV infusion over an hour
  Arms: TB006
Drug: Placebo — Normal saline administered through IV infusion over an hour
  Arms: Placebo

SUMMARY:
This multi-center, randomized, parallel-group, double-blind, placebo-controlled study will evaluate the efficacy and safety of TB006 in participants with an Acute Ischemic Stroke (AIS) event with 57 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 40 kilograms per meters squared (kg/m^2), inclusive
* Clinical diagnosis of AIS in anterior circulation, supported by evidence of a new stroke on acute brain computed tomography (CT) or magnetic resonance imaging (MRI) consistent with the clinical diagnosis.
* Able to be randomized and dosed within 7 days of index stroke event. The last known awake time will be used for participants whose stoke occurred during sleep.
* National Institute of Health Stroke Scale total score of 7 to 21, inclusive
* Participants may have received standard of care therapy including recombinant tissue plasminogen activator (r-tPA), thrombectomy, mannitol, hypertonic saline, and other treatments per local guidelines as determined by the Investigator. Participants who have received r-tPA within the first day of their stroke event are eligible. However, study drug administration must begin more than 24 hours following r-tPA administration.

Exclusion Criteria:

* Evidence of severe stroke on imaging (e.g., sulcal effacement or blurring of gray-white junction in greater than 1/3 of middle cerebral artery [MCA] territory, Alberta Stroke Program Early CT [ASPECT] score of 0 to 4 based on head CT, acute infarct volume on MRI diffusion weighed imaging ≥70 mL based on acute imaging studies performed under the standard of care
* Lacunar or isolated brainstem or cerebellar stroke based on clinical assessment and available acute imaging studies performed under the standard of care
* Evidence of seizure at the onset of index stroke
* Evidence of acute myocardial infarction (MI) at Baseline, including any of the following:

  1. Acute ST elevation MI;
  2. Acute decompensated heart failure, or New York Heart Association Class III/IV heart failure;
  3. Admission for an acute coronary syndrome, MI, cardiac arrest, or non-voluntary coronary intervention (percutaneous coronary intervention or coronary artery surgery) within the past 3 months.
  4. QT interval corrected using Bazett's formula (QTcB) >520 milliseconds (msec).
* Evidence of acute intracranial or subarachnoid hemorrhage or evidence of active bleeding based on acute brain CT or MRI performed under the standard of care. However, petechial hemorrhages of ≤ 1 centimeter (cm) are not exclusionary.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Recovery Success Measured by modified Rankin Scale (mRS) score of 0-1 on the final mRS assessment. | Day 90
  The Modified Rankin Scale (mRS) measures neurological disability or dependence of participants with stroke on a scale of 0 to 6 and scores indicate the following: 0 - No symptoms; 1 - No significant disability; 2 - Slight disability; 3 - Moderate disability; 4 - Moderately severe disability; 5 - Severe disability; 6 - Dead. Higher score indicates worse condition.

SECONDARY OUTCOMES:
Percentage of Participants with Clinically Significant Improvement on the National Institutes of Health Stroke Scale (NIHSS) | At Days 29, 57 and 85
  Clinically significant improvement is defined as a 4-point decrease on the NIHSS
Change from Baseline in Neurological Function on the NIHSS | Baseline and through Day 85
  The NIHSS is composed of 11 items, each of which rates a specific parameter of ability or function. Each item is rated on a scale of 0 to 4. A score of 0 indicates normal function, with higher scores indicating greater degree of impairment. The individual item scores are added to calculate the NIHSS total score. The minimum score being a 0 (no impairment) and maximum possible score is 42 (death). Higher scores indicate worse condition.
Percentage of Participants with Clinically Significant Improvement on the mRS | At Days 29, 57 and 85
  Clinically Significant Improvement is defined as 1-point decrease on the mRS
Change from Baseline in the Montreal Cognitive Assessment (MoCA) Total Score | Baseline and at Days 29, 57, and 85
  The MoCA is a brief screening instrument designed to assess mild cognitive impairment in a variety of participant conditions. The MoCA assesses eight cognitive domains: visuospatial ability, executive function, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space. Scores on the MoCA range from 0 to 30, with lower scores indicating greater impairment.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 141
Number of Participants with Clinically Significant Clinical Laboratory Parameter Values | Up to Day 141
Number of Participants with Clinically Significant Vital Sign Values | Up to Day 141
Number of Participants with Clinically Significant 12-Lead Electrocardiogram Findings | Up to Day 141
Number of participants with Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Day 141
  The C-SSRS is a suicidal ideation and behavior rating scale with yes/no responses. For each of the 5 items of the C-SSRS related to suicidal ideation intensity, an individual's degree of suicidal ideation is rated on a 0-5 scale with 0: no suicidal behavior and 5: active suicidal ideation. The total score is the sum of the 5 intensity item scores (total score ranges from 0 to 25). Higher scores in the scale indicate greater disease severity.
Number of Participants with Clinically Significant Physical Examination Findings | Up to Day 141
Number of Participants with Anti-drug Antibodies | Up to Day 141
Plasma concentration of TB006 | Pre-dose and post-dose on Days 1, 29, 57, 85 and 141

CONTACTS AND LOCATIONS:
Overall Officials: TrueBinding, Inc., Study Director — TrueBinding, Inc.

IPD SHARING:
Plan to Share IPD: No